CLINICAL TRIAL: NCT04009343
Title: Field Study of the Pharmacokinetics and Pharmacodynamics of Artemisinin-based Combination Therapy for Gametocyte Clearance and Post-treatment Chemoprotection in Zambian Children With Uncomplicated Falciparum Malaria
Brief Title: Pharmacokinetics and Pharmacodynamics of the Gametocytocidal and Post-treatment Chemoprotective Effects of Antimalarials
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Tropical Diseases Research Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00007663
Record Dates: First submitted 2019-06-07; First posted 2019-07-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Uncomplicated Falciparum Malaria
MeSH Terms: interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and clinical trial nurses and pharmacists will be aware of the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Artemether-lumefantrine (Active Comparator): Standard 6-dose regimen
  Interventions: Drug: Artemether-lumefantrine
- Dihydroartemisinin-piperaquine (Experimental): Standard 3-dose regimen
  Interventions: Drug: Dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: Artemether-lumefantrine — Children will receive artemether-lumefantrine (20/120 mg) dosed according to weight (5 to <15 kg: 1 tablet, 15 to <25 kg: 2 tablets) at 0, 8, 24, 36, 48 and 60 hours. Medications will be administered according to the manufacturer's instructions.
  Other Names: Coartem®
  Arms: Artemether-lumefantrine
Drug: Dihydroartemisinin-piperaquine — Children will receive dihydroartemisinin-piperaquine (40/320 mg) dosed according to weight (5 to <8 kg: 1/2 tablet, 8 to <11 kg: 3/4 tablet, 11 to <17 kg: 1 tablet, 17 to <25 kg: 1 1/2 tablets) at 0, 24, and 48 hours. Medications will be administered according to the manufacturer's instructions.
  Other Names: D-Artepp®
  Arms: Dihydroartemisinin-piperaquine

SUMMARY:
Single-center phase II/III clinical investigation of the pharmacokinetics and pharmacodynamics of artemether-lumefantrine and dihydroartemisinin-piperaquine for gametocyte clearance and post-treatment chemoprotection in Zambian children with uncomplicated falciparum malaria.

DETAILED DESCRIPTION:
Artemisinin-based combination therapies (ACTs) are the first-line agents for uncomplicated falciparum malaria. Artemether-lumefantrine (AL) is the most widely adopted ACT in sub-Saharan Africa for case management. Dihydroartemisinin-piperaquine (DP) is increasingly used for mass drug administration in malaria eliminating regions, and is being explored as a candidate for intermittent preventive therapy. AL and DP possess similar clinical efficacy against uncomplicated falciparum malaria in areas of drug susceptible parasites. However, AL appears to clear gametocytes (the transmissible stage of the malaria parasite) more rapidly than DP, while DP confers a longer duration of post-treatment protection against reinfection. It is not known whether the observed difference in gametocyte clearance between AL and DP is due to pharmacokinetic (PK) and/or pharmacodynamic (PD) differences of the artemisinin derivatives, PK/PD features of the non-artemisinin companions, or contributions from both. The longer duration of protection against reinfection provided by DP is due to the long elimination half-life of the partner drug, but further characterization of its relative benefit in high-transmission settings compared to AL is needed to inform malaria drug policy. The investigators are conducting a single-center randomized controlled clinical trial comparing the efficacies of AL and DP for gametocyte clearance and post-treatment chemoprotection among 6- to 59-month-old children with uncomplicated falciparum malaria in a high malaria transmission area of northern Zambia. Children with microscopy-confirmed Plasmodium falciparum monoinfection will be admitted for 72 hours for directly observed therapy with either AL or DP and serial sampling for parasite clearance and multi-dose PK measurements. Twenty children from each arm will be recruited to an intensive PK subgroup. Participants will be followed for 9 weeks for outcome assessment according to World Health Organization-defined clinical endpoints and to measure clearance of the long-acting partner drugs. Parasite genotyping will be done to distinguish recrudescence from reinfection and query genetic markers of drug resistance. Participants will contribute fecal specimens to help investigate bidirectional associations between the intestinal microbiota and antimalarial drug pharmacokinetics, as well as enterotype association with risk of reinfection.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥10 kg
* Any indication for malaria diagnostic testing as determined by a treating provider (e.g., fever or history of fever)
* P. falciparum parasitemia (by microscopy) of any density not meeting criteria for severe malaria
* Ability to swallow oral medication
* Ability and willingness of parents or guardians to comply with study protocol for the duration of the study and to comply with the study follow-up visit schedule
* Residence within hospital catchment area
* Signed informed consent obtained from a legal representative of the participant

Exclusion Criteria:

* Complicated or severe falciparum malaria as defined by WHO criteria
* Hemoglobin concentration < 7 g/dL
* Use of any drug with antimalarial activity within the prior 4 weeks
* History of hypersensitivity reaction or intolerance to AL or DP
* Co-infection with Plasmodium spp. other than P. falciparum as determined by microscopy
* Confirmed or suspected concurrent acute infection other than malaria (e.g. measles, acute lower respiratory tract infection)
* Current therapy with QT interval-prolonging agents
* Family history of sudden cardiac death or personal history of cardiac disease
* Residence outside the study area, or plan to leave the study area
* Residence in foster care or otherwise under government supervision
* Previous enrollment in the study, or enrollment in any other investigational drug trial during the previous 30 days
* Presence of any other condition or abnormality that in the opinion of the investigator would compromise the safety of the participant or the quality of the data

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Treatment outcome | 9 weeks
  Defined according to World Health Organization (WHO) classification as adequate clinical and parasitological response, early treatment failure, late clinical failure, or late parasitological failure corrected by genotyping to distinguish reinfection from recrudescent infection.
Area-under-the-curve (AUC) of the gametocyte concentration-time curve | 72 hours
  Primary gametocyte-related pharmacodynamic (PD) endpoint of the study
Incidence of reinfection during the 9-week follow-up period | 9 weeks
  Primary measure of the post-treatment chemoprotective effect of the drugs

SECONDARY OUTCOMES:
Elimination half-life of the gametocyte concentration-time curve | 72 hours up to 9 weeks for those with persistent gametocytemia
  Alternative PD outcome of gametocyte dynamics
Change over time of the gametocyte sex ratio (female:male) | 72 hours up to 9 weeks for those with persistent, emergent, or recurrent gametocytes
  The ratio of female and male gametocytes over time during treatment is a hypothesized marker of transmissibility
Elimination half-life of the asexual parasite concentration-time curve | 72 hours
  In addition to gametocyte dynamics, asexual parasite dynamics and how they relate to PK parameters and other covariates with also be examined
Allele frequency of genetic markers of parasite drug resistance in initial vs. recurrent parasites and fast vs. slow clearing parasites | 9 weeks
  Relative barriers to drug resistance of AL and DP will be tested using known and newly described parasite genetic markers of resistance and association with phenotypic susceptibility
Incidence of treatment-emergent adverse events (safety and tolerability) | 9 weeks
  We will assess adverse events and serious adverse events associated with the study drugs in accordance with the WHO Toxicity Grading Scale for Determining the Severity of Adverse Events

OTHER OUTCOMES:
AUC of the plasma concentration-time curve | 72 hours (artemisinin derivatives) and 9 weeks (long-acting companions)
  Pharmacokinetic (PK) endpoint of the study, determined for each drug and drug metabolite
Peak plasma concentration (Cmax) of study drugs and metabolites | 72 hours (artemisinin derivatives) and 9 weeks (long-acting companions)
  PK endpoint of the study, determined for each drug and drug metabolite
Oral clearance (Cl/F) for all drug analytes | 72 hours (artemisinin derivatives) and 9 weeks (long-acting companions)
  PK endpoint of the study, determined for each drug and drug metabolite
Nutrition status-related associations with drug PK | 72 hours (artemisinin derivatives) and 9 weeks (long-acting companions)
  In nonlinear mixed effects PK models, we will test associations between nutrition status (weight-for-age Z score) and drug PK parameters
Body surface area-related associations with drug PK | 72 hours (artemisinin derivatives) and 9 weeks (long-acting companions)
  We will test, in nonlinear mixed effects PK models, associations between body surface area and drug PK
Gut microbiota enterotype | 9 weeks
  We will characterize the gut microbiota of study participants and examine bidirectional associations between enterotype and drug PK, and enterotype and incidence of reinfection

CONTACTS AND LOCATIONS:
Overall Officials: William J Moss, MD MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Tropical Diseases Research Centre, Ndola, Copperbelt, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available to other researchers upon reasonable request. Parasite clearance and drug resistance data will be contributed to the Worldwide Antimalarial Resistance Network database.

DOCUMENTS (1):
  • Informed Consent Form (2019-05-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT04009343/ICF_001.pdf